CLINICAL TRIAL: NCT01245907
Title: Climacteric Therapy With Applied Relaxation Using InterNet - CARIN Study
Brief Title: Climacteric Therapy With Applied Relaxation Using InterNet
Acronym: CARIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unacceptable high drop-out rate.
Sponsor: Mats Hammar (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Mats Hammar, Professor, Ostergotland County Council, Sweden
Organization: Ostergotland County Council, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100528/CARIN
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Hot Flashes; Menopause
Keywords: Hot flashes; Menopause; HRQoL; Applied relaxation; Insomnia; Women's knowledge
MeSH Terms: conditions — Hot Flashes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Applied relaxation (Experimental): Applied relaxation given by Internet during 10 weeks as a number of text-documents, audio-files and e-mail mediated support from therapists
  Interventions: Behavioral: Applied relaxation
- Waiting-list/control (No Intervention): No intervention for 10 weeks but the same registrations and diaries and forms as the interventional group

INTERVENTIONS:
Behavioral: Applied relaxation — Applied relaxation given by Internet during 10 weeks as a number of text-documents, audio-files and e-mail mediated support from therapists
  Arms: Applied relaxation

SUMMARY:
The aim is to evaluate effects of internet-based applied relaxation (a simplified version of cognitive behavioral therapy) for women with menopausal symptoms mainly vasomotoric symptom (VMS), i.e. hot flashes and sweating. Sixty postmenopausal women with VMS will be recruited and 30 randomized to applied relaxation (AR) via internet and 30 to a control group which is a non-treated waitlist group.

At baseline, after 10 weeks of therapy and six, 12 and 24 months after end of therapy women will be asked to fill in diaries about hot flashes and answer questionnaires on Quality of Life (Women's Health Questionnaire; WHQ, anxiety and depression measured with Hospital Anxiety and Depression Scale; HADS and one measuring sleep, Insomnia Severity Index; ISI as well as one about knowledge of the climacteric and hormone therapy).

The waiting list group will be offered internet based AR after 10 weeks with the same follow-up as the treatment group.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 7 moderate or severe hot flashes per 24 h or 50 hot flashes per week in average at least during one week before randomization (mild = hot flash without sweating as recognized by the woman but not disturbing the woman, moderate = hot flash and sweating as recognized by the woman but that does not lead to disruption of ongoing activity, severe = hot flash with sweating that leads to disruption of ongoing activity)
* Natural menopause (at least 12 months without any menstrual bleedings at all)
* At least 45 years of age during present year
* Access to computer with Internet
* Ability to read and speak Swedish
* Freely informed concent for participation

Exclusion Criteria:

* Induced menopause (e.g. hysterectomy, oophorectomy, chemotherapy, radiation therapy over abdominal- and/or pelvic region)
* Early or premature menopause (before 45 years of age)
* Breastcancer disease with ongoing therapy with antiestrogen or aromatase inhibitors
* Ongoing usage or use during the last month of hormone therapy or other treatment aimed for hot flashes (e.g. natural remedies affecting hot flashes, acupuncture, dietary supplements aimed to treat hot flashes
* Treatment with psychopharmacological drugs (e.g SSRI or SNRI) or frequent use of benzodiazepines, drugs for insomnia(> 1 times/week)
* Untreated or unstable endocrinological- or metabolic disease( e.g thyroid disease)
* Undiagnosed vaginal bleeding after menopause

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in numbers of hot flashes per 24 h | Baseline to 10 weeks of treatment/control group
  Numbers of hot flashes per 24 h daily recorded in hot flash diary from baseline throughout 10 weeks of treatment. Comparison between treatment group and control group (waitlist)

SECONDARY OUTCOMES:
Health related Quality of life (HRQoL) | Baseline to 10 weeks of treatment/control group
  HRQoL measured with WHQ at baseline and after 10 weeks. Comparison between treatment group and control group (waitlist)
Severity of insomnia | Baseline to 10 weeks of tratment/control group
  Insomnia measured with Insomnia severity Index (ISI)at baseline and after 10 weeks. Comparison between treatment group and control group (waitlist)
Women's knowledge about menopause and treatment of menopausal related symptoms | Baseline to 10 weeks of treatment/control group
  Knowledge measured with a questionnaire measuring women's knowledge about menopause and treatment of menopausal related symptoms at 10 baseline and after 10 weeks. Comparison between the treatment group and the control group (waitlist)
Change in numbers of hot flashes per 24 h, WHQ, ISI | Baseline to 6, 12 and 24 months after end treat treatment
  Assessment if changes from baseline to 10 weeks persist after 6, 12 and 24 months after end of treatment in the treatment group.
Adverse Event | Baseline to 10 weeks of treatment/control group
  Open ended questions about occurence of adverse events during the treatment period. Comparison between the treatment group and the control group (waitlist)

CONTACTS AND LOCATIONS:
Overall Officials: Mats L Hammar, MD, Principal Investigator — Linkoeping University
Locations (1):
- County Council of Östergötland, Kvinnokliniken, Linköping, Sweden

REFERENCES:
- [Background] Nedstrand E, Wyon Y, Hammar M, Wijma K. Psychological well-being improves in women with breast cancer after treatment with applied relaxation or electro-acupuncture for vasomotor symptom. J Psychosom Obstet Gynaecol. 2006 Dec;27(4):193-9. doi: 10.1080/01674820600724797. PMID 17225620
- [Background] Nedstrand E, Wijma K, Wyon Y, Hammar M. Applied relaxation and oral estradiol treatment of vasomotor symptoms in postmenopausal women. Maturitas. 2005 Jun 16;51(2):154-62. doi: 10.1016/j.maturitas.2004.05.017. PMID 15917156
- [Background] Ost LG. Applied relaxation: description of a coping technique and review of controlled studies. Behav Res Ther. 1987;25(5):397-409. doi: 10.1016/0005-7967(87)90017-9. No abstract available. PMID 3318800
- [Background] Carlbring P, Ekselius L, Andersson G. Treatment of panic disorder via the Internet: a randomized trial of CBT vs. applied relaxation. J Behav Ther Exp Psychiatry. 2003 Jun;34(2):129-40. doi: 10.1016/s0005-7916(03)00026-0. PMID 12899896
- [Background] Furmark T, Carlbring P, Hedman E, Sonnenstein A, Clevberger P, Bohman B, Eriksson A, Hallen A, Frykman M, Holmstrom A, Sparthan E, Tillfors M, Ihrfelt EN, Spak M, Eriksson A, Ekselius L, Andersson G. Guided and unguided self-help for social anxiety disorder: randomised controlled trial. Br J Psychiatry. 2009 Nov;195(5):440-7. doi: 10.1192/bjp.bp.108.060996. PMID 19880935
- [Background] Lindh-Astrand L, Brynhildsen J, Hoffmann M, Kjellgren KI, Hammar M. Knowledge of reproductive physiology and hormone therapy in 53- to 54-year-old Swedish women: a population-based study. Menopause. 2007 Nov-Dec;14(6):1039-46. doi: 10.1097/gme.0b013e31803816ca. PMID 17519805
- [Background] Wiklund I, Karlberg J, Lindgren R, Sandin K, Mattsson LA. A Swedish version of the Women's Health Questionnaire. A measure of postmenopausal complaints. Acta Obstet Gynecol Scand. 1993 Nov;72(8):648-55. doi: 10.3109/00016349309021159. PMID 8259753
- [Background] Lisspers J, Nygren A, Soderman E. Hospital Anxiety and Depression Scale (HAD): some psychometric data for a Swedish sample. Acta Psychiatr Scand. 1997 Oct;96(4):281-6. doi: 10.1111/j.1600-0447.1997.tb10164.x. PMID 9350957
- [Background] Karling P, Hammar M, Varenhorst E. Prevalence and duration of hot flushes after surgical or medical castration in men with prostatic carcinoma. J Urol. 1994 Oct;152(4):1170-3. doi: 10.1016/s0022-5347(17)32530-2. PMID 8072086
- [Background] Holmberg L, Iversen OE, Rudenstam CM, Hammar M, Kumpulainen E, Jaskiewicz J, Jassem J, Dobaczewska D, Fjosne HE, Peralta O, Arriagada R, Holmqvist M, Maenpaa J; HABITS Study Group. Increased risk of recurrence after hormone replacement therapy in breast cancer survivors. J Natl Cancer Inst. 2008 Apr 2;100(7):475-82. doi: 10.1093/jnci/djn058. Epub 2008 Mar 25. PMID 18364505
- [Background] Berg G, Gottwall T, Hammar M, Lindgren R. Climacteric symptoms among women aged 60-62 in Linkoping, Sweden, in 1986. Maturitas. 1988 Oct;10(3):193-9. doi: 10.1016/0378-5122(88)90022-9. PMID 3185293
- [Background] Hoffmann M, Hammar M, Kjellgren KI, Lindh-Astrand L, Brynhildsen J. Changes in women's attitudes towards and use of hormone therapy after HERS and WHI. Maturitas. 2005 Sep 16;52(1):11-7. doi: 10.1016/j.maturitas.2005.06.003. PMID 16023804
- [Derived] Lindh-Astrand L, Holm AC, Sydsjo G, Andersson G, Carlbring P, Nedstrand E. Internet-delivered applied relaxation for vasomotor symptoms in postmenopausal women: lessons from a failed trial. Maturitas. 2015 Apr;80(4):432-4. doi: 10.1016/j.maturitas.2015.01.010. Epub 2015 Feb 2. PMID 25700856